## Train-of-four monitoring using the Tetragraph® Neuromuscular Transmission Monitor: Tolerance to preoperative electrode placement

NCT05964166

May 16, 2023

**Statistical Analysis** 

## Statistical analysis

Statistical analysis was conducted using SAS 9.4. To assess the normality of continuous variables, the Shapiro-Wilk test was employed. Given the skewed distribution of the data, continuous variables were presented using median and interquartile ranges (IQR). Categorical variables were reported as frequency and percentages. Non-parametric data including the Likert score ratings were summarized and presented using median and IQRs. To analyze the data statistically, a Wilcoxon sum-rank test was performed for between group comparisons of continuous variables while a Chi-square test was utilized to investigate associations among categorical variables. Furthermore, a binary logistic regression analysis was conducted to evaluate the relationship between age and the odds of keeping the sensor intact before entering the OR. A significance level of P < 0.05 was applied for all statistical tests.